CLINICAL TRIAL: NCT00748137
Title: Bolus Insulin Card Calculator Randomised Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: John Hunter Children's Hospital (Other)
Collaborators: Royal North Shore Hospital (Other); Sydney Children's Hospitals Network (Other); Royal Children's Hospital (Other); Lady Cilento Children's Hospital, Brisbane (Other); NovoNordisk Pharmaceuticals (Unknown)
Responsible Party: Dr Donald Anderson, Staff Specialist, John HUnter Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/04/26/5.01
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2009-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Youth; Insulin dose
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed dose (Active Comparator): Fixed meal size and fixed aspart insulin dose except for minor changes based on measured blood glucose. Detemir basal insulin.
  Interventions: Other: Fixed dose
- ezy-BICC dose calculation card (Experimental): variable meal size with variable aspart insulin dose determined with use of individualised dose calculation card. Detemir basal insulin.
  Interventions: Device: ezy-BICC dose calculation card

INTERVENTIONS:
Device: ezy-BICC dose calculation card — small laminated table lists the dose of insulin to administer based on BGL and carbohydrate to be consumed - individualised for each study subject
  Arms: ezy-BICC dose calculation card
Other: Fixed dose — Approach where study subject is prescribed a set amount of carbohydrate to eat each meal and set dose of rapid acting insulin. Minor modifications may be made if the measured BGL is out of target
  Arms: Fixed dose

SUMMARY:
In pediatric patients with type 1 diabetes using subcutaneous injections; a randomised controlled trial comparing the effects of fixed carbohydrate exchanges and insulin doses to the use of variable size meals and insulin doses determined with a bolus insulin calculation card.

ELIGIBILITY:
Inclusion Criteria:

* Age 11 - 18 years old
* Currently using indvidual subcutaneous injections (not CSII)

Exclusion Criteria:

* HbA1c > 9.5%
* Serious illness

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-10 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
24 hours BGL > 8.3mmol/l (CGMS) | 3 months

SECONDARY OUTCOMES:
HbA1c | 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Gosford District Hospital, Gosford, New South Wales
  - John Hunter Children's Hospital, Newcastle, New South Wales
  - Sydney Children's Hospital, Sydney, New South Wales
  - Mater Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Brisbane, Queensland